CLINICAL TRIAL: NCT05537012
Title: Incidence of Unresectable Cases of Cervical Cancer in Gyne-oncology Unit of Alexandria University Hospital and Its Relation to Pathological Types, Grading and Lymph Vascular Space Invasion
Brief Title: Incidence of Unresectable Cases of Cervical Cancer
Status: Completed | Type: Observational
Sponsor: HOSSAM ALSUKARI (Other)
Responsible Party: Sponsor-Investigator, HOSSAM ALSUKARI, Associate professor, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: SOKKARY10
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: clinical and radiological staging, pathological types, grading and lymphovascular space invasion — 70 cases of cervical cancer diagnosed by biopsy taking and histopathological examination will be included in the study, clinicoradiological staging was done to all cases to calculate the incidence of unresectable cases and to indentify its relation to pathological types, grading and lymph vascular space invasion.

SUMMARY:
Objective : to calculate the incidence of unresectable cases of cervical cancer in gyne-oncology unit of Alexandria university hospital and to indentify its relation to pathological types, grading and lymph vascular space invasion.

Patients and methods: 70 cases of cervical cancer diagnosed by biopsy taking and histopathological examination will be included in the study, clinicoradiological staging was done to all cases to calculate the incidence of unresectable cases and to indentify its relation to pathological types, grading and lymph vascular space invasion

ELIGIBILITY:
Inclusion Criteria:

* cervical cancer

Exclusion Criteria: none

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: random cases of cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
clinical and radiological staging | 10 days
  70 cases of cervical cancer diagnosed by biopsy taking and histopathological examination will be included in the study, clinicoradiological staging was done to all cases to calculate the incidence of unresectable cases and to indentify its relation to pathological types, grading and lymph vascular space invasion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hossam Hassan El Sokkary, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided